CLINICAL TRIAL: NCT02114255
Title: The Effects of BCG-vaccination on the Immune Response Induced by Influenza-vaccination in Healthy Volunteers. A Pilot Proof-of-principle Study.
Brief Title: Effects of BCG on Influenza Induced Immune Response
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BCG_influenza
Record Dates: First submitted 2014-03-10; First posted 2014-04-15 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Influenza Virus Infection; Trained Immunity
Keywords: Influenza; Trained immunity; BCG
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCG vaccination (Experimental): BCG vaccination
  Interventions: Biological: BCG
- NaCl 0.9% (Placebo Comparator): administration of NaCl 0.9%.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Administration of 0.9% NaCl.
  Arms: NaCl 0.9%
Biological: BCG — Vaccination with the live attenuated BCG vaccine.
  Arms: BCG vaccination

SUMMARY:
In the present study, the investigators want to investigate whether prior BCG-vaccination improves the efficacy of influenza ("the flu") vaccination in young and/or old healthy volunteers and consequently could protect against influenza virus infection.

DETAILED DESCRIPTION:
Influenza virus infection leads to millions of cases of severe illnesses worldwide and up to an estimated 500.000 deaths annually. The potential for the sudden emergence of pandemic influenza strains represents an incessant threat on even a larger scale. seasonal influenza vaccination is the backbone of influenza management. However, antibodies generated by vaccination, most often do not effectively neutralize emergent strains due to the high mutation rate of the influenza viral genome. In addition, although vaccination is effective in up to 85% of healthy adults, only 40-60% of the elderly are able to mount an protective antibody response due to an agerelated decline in immune function (so-called immunoscenescence). As a result, the protective effects of influenza vaccination are limited, and strategies to improve host immune defenses against influenza virus infection per se, and following influenza vaccination, are highly warranted.

It is suggested that prior vaccination with Bacille Calmette-Guérin (BCG) could enhance resistance to other infectious diseases in addition to protection to tuberculosis (TBC) and, in mice, protection of prior BCGvaccination against influenza infection was demonstrated long ago. However, only recently substantial evidence for these nonspecific beneficial effects of BCG-vaccination in humans has been provided by several randomized clinical trials. Considering these potentiating effects of BCG-vaccination, it could be a viable strategy to improve efficacy of influenza vaccination, and/or enhance immune defenses against influenza virus infection per se. If so, this would have an enormous impact on clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤35 yrs
* Male
* Healthy

Exclusion Criteria:

* History of influenza vaccination within the year prior to study entry
* History of BCG vaccination within 5 years prior to study entry
* History of Mantoux testing within the year prior to study entry
* Vaccination other than BCG or influenza, within 3 months prior to study or within study period
* Medical history of any disease associated with immune deficiency
* Clinically significant acute illness, including infections, within 4 weeks before vaccination
* Participation in a drug trial or donation of blood 3 months prior to study entry
* Use of recreational drugs within 21 days prior to experiment day
* Recent hospital admission or surgery with general anaesthesia (<3 months)
* Known chronic kidney or liver disease
* Latent or active tuberculosis infection

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Difference in influenza antibody titres between BCG-vaccinated subjects and subjects in the control group | Day 14, day 21, day 28, day 42 (±2 days)
Difference in Thrombocyte function between BCG-vaccinated subjects and subjects in the control group | Day 0, day 14, day 21, day 28, day 42 (±2 days)

SECONDARY OUTCOMES:
Proportion of participants in each group who achieved seroprotection (defined by antibody titre ≥1:40). | day 21, day 28, day 42 (±2 days)
Proportion of participants in each group who achieved seroconversion (defined by a ≥4-fold rise in antibody titre). | day 21, day 28, day 42 (±2 days)
IFN-gamma/IL-10 production of leukocytes ex vivo stimulated with inactivated/live influenza virus (0.1ug HA/ml). | Day 0, day 14, day 28, day 42 (±2 days)
Production of Type 1 IFNs, IL-17 and IL-22 by leukocytes ex vivo stimulated with inactivated/live influenza virus (0.1ug HA/ml). | Day 0, day 14, day 28, day 42 (±2 days)
Production of other inflammatory mediators (including TNFα, IL-1β, IFN-gamma, IL-10, IL-17, IL-22) by leukocytes ex vivo stimulated with different not-related stimuli (including m. tuberculosis, s. aureus, c. albicans, and inactivated influenza). | Day 0, day 21, day 28, day 42 (±2 days)
Inflammatory transcriptional pathways (by use of qPCR/microarrays) . | Day 0, day 14, day 28, day 42 (±2 days)
Granzyme B production of leukocytes ex vivo stimulated with inactivated/live influenza virus (0.1ug HA/ml). | Day 0, day 14, day 28, day 42 (±2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, The Netherlands
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands